CLINICAL TRIAL: NCT00001218
Title: Development of Normative Ultrasound Databases of Tongue Surface Configuration
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 870016; 87-CC-0016
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-01

CONDITIONS: Healthy; Speech Disorders
Keywords: Baseline Data; Curve Averaging; Curve Fitting; Movement Patterns; Normative Data; Polar Distribution; Tongue; Tongue Shape; Ultrasound
MeSH Terms: conditions — Speech Disorders

SUMMARY:
Our past ultrasound research has indicated a need for baseline normative tongue data against which to compare our disordered speech populations. Subjects with normal speech and hearing who represent different ages and sexes, will be studied with respect to tongue shape and movement patterns. Recently developed parameters such as curve fitting, curve averaging, and polar coordinates will be used to create baseline data categories. In addition, new parameters and improved instruments will be developed as previously to produce a data base which can be used across disciplines.

DETAILED DESCRIPTION:
Our past ultrasound research has indicated a need for baseline normative tongue data against which to compare our disordered speech populations. Subjects with normal speech and hearing who represent different ages and sexes, will be studied with respect to tongue shape and movement patterns. Recently developed parameters such as curve fitting, curve averaging, and polar coordinates will be used to create baseline data categories. In addition, new parameters and improved instruments will be developed as previously to produce a data base which can be used across disciplines.

ELIGIBILITY:
Healthy normal subjects.

No reconstructive tongue surgery.

No radiation for head and neck malignancy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 1987-02; Study Completion 2001-01

CONTACTS AND LOCATIONS:
Locations (1):
- Warren G. Magnuson Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Sonies BC, Wang C, Sapper DJ. Evaluation of normal and abnormal hyoid bone movement during swallowing by use of ultrasound duplex-Doppler imaging. Ultrasound Med Biol. 1996;22(9):1169-75. doi: 10.1016/s0301-5629(96)00158-5. PMID 9123641